CLINICAL TRIAL: NCT02350855
Title: To Study the Impact of Nutritional Intervention in Delaying the Progression of Cachexia to Refractory Cachexia in Female Cancer Patients: A Study Based in India
Brief Title: Impact of Nutritional Intervention in Indian Female Cancer Cachexia Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Neha Kapoor, Research Scholar, University of Westminster
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12_13_11
Record Dates: First submitted 2015-01-26; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Cachexia; Cancer
Keywords: Nutrition intervention; Palliative care; Public Health; Quality of life; Tailored food formula; Body weight
MeSH Terms: conditions — Cachexia; Neoplasms; Body Weight | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Patients in the intervention group were given dietary supplement (Improved Atta: 100 g) daily along with nutritional counseling and physical activity counseling for six months.
  Interventions: Dietary Supplement: Improved Atta; Other: Nutritional counseling; Behavioral: Physical activity counseling
- Control group (Other): Patients in the control group were given nutritional and physical activity counseling for six months every fortnight.
  Interventions: Other: Nutritional counseling; Behavioral: Physical activity counseling

INTERVENTIONS:
Dietary Supplement: Improved Atta — Improved Atta is a multi macro- micronutrient bread mix. Patients were given 100 grams of Improved Atta (in the from of unleavened bread) everyday for consumption for six months.
  Arms: Intervention group
Other: Nutritional counseling — Dietary counseling for 30 minutes was imparted to all patients on every hospital visits by the researcher. Consumption of cereals, roots and tubers, vegetables, legumes, nuts, energy dense fruits, milk products (and eggs for non-vegetarians) was encouraged in their daily diets.
Behavioral: Physical activity counseling — Depending on the physical status of the patients, low level of physical activity (walking and/or stairs), was encouraged daily during counseling sessions.

SUMMARY:
The main aim of the study is to assess the effectiveness of tailored nutritional intervention in delaying the progression of cachexia to refractory cachexia in adult female cancer patients.

The tested hypothesis stated that intake of nutrient rich bread mix (along with dietary and physical activity counselling) for six months, improved the anthropometric and biochemical indices in free-living patients suffering from cancer cachexia.

DETAILED DESCRIPTION:
Patients were randomly distributed into two groups i.e. control and intervention group. 30 patients were allocated in intervention group and received nutrient rich bread mix i.e. IAtta (100 g) along with dietary and physical activity counseling and 33 patients were allocated in the control group who received only dietary and physical activity counseling. Patients in the intervention group collected 14 packets of 100 g of IAtta every fortnight during their clinician appointments while the control patients were advised regarding their dietary habits at every clinician visit for 6 months.

Dietary counseling for 30 minutes was imparted to all patients on each visit by the researcher. Depending on the physical status of the patients, low level of physical activity (walking and/or stairs), was encouraged daily during counseling sessions.

Nutritional, biochemical, quality of life and anthropometric estimations were assessed at baseline, after 3 months and at 6 months of intervention for all patients.

Patients' daily energy, carbohydrate, protein and fat intake were calculated using food frequency (Indian Migrant study food frequency questionnaire- IMS-FFQ) questionnaire and two day 24 hour recall data. PG-SGA questionnaire was used to monitor patient nutritional status throughout the study.

EORTC-QLQ- C30 questionnaire was used to analyse patients' quality of life and asked personally by the researcher.

Haemoglobin and serum albumin levels were assessed at the start of the study, after 3 months and at 6 months of intervention for all patients.

Indian Migrant Study Physical Activity questionnaire (IMS-PAQ) was used to assess patients' physical activity throughout the day.

Anthropometric estimations included body weight, mid upper arm circumference and four site skin fold thickness (SFT) measurement (i.e. triceps, biceps, subscapular and suprailiac).

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years and above.
* Diagnosed with cancer.
* Weight loss >5% from pre-treatment weight or BMI<20kg/m2.
* Hemoglobin level <12 g/dl.
* Energy intake < 1500 kcal/d (to be assessed on consultation).

Exclusion Criteria:

* Incapable to provide written consent.
* Patient diagnosed with refractory cachexia.
* Life expectancy < 3 months.
* Unresponsive to anti-cancer therapy.
* Patient is a pregnant woman or a nursing mother.
* Suffering from secondary illnesses.
* Gastrointestinal tract defects which affect nutrient absorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-12; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Body weight | 6 months
  Body weight was assessed using a Tanita segmental composition scale at baseline, mid-intervention (3 months) and at the end of intervention (6 months).

SECONDARY OUTCOMES:
Mid upper arm circumference (MUAC) | 6 months
  MUAC was measured using a non-stretchable measuring tape at baseline, mid-intervention (3 months) and at the end of intervention (6 months).
Body fat percentage (BF%) | 6 months
  Four site skin fold thickness (SFT) measurement (i.e. triceps, biceps, subscapular and suprailiac) by the help of scientific Harpenden Skinfold Caliper was noted to the nearest 0.2mm reading, to calculate percentage body density. Body fat percentage was calculated using body density value in Siri equation. SFT was measured at baseline, mid-intervention (3 months) and end of intervention (6 months) to determine the BF%.
Nutritional status assessment (Indian Migrant study food frequency questionnaire (IMS-FFQ), two day 24 hour dietary recall and patient generated subjective global assessment) | 6 months
  Indian Migrant study food frequency questionnaire (IMS-FFQ), two day 24 hour dietary recall and patient generated subjective global assessment were used to assess patient nutritional status at baseline, mid-intervention and end of intervention (6 months).
  Food frequency questionnaire and 24 hour dietary recall is an accurate method to record the frequency of consumption of individual foods and can help provide information on patients' eating patterns.IMS-FFQ consists of 184 commonly consumed food items and was validated among the rural and urban Indian population. PG-SGA is most effective and sensitive tool for assessing and evaluating cancer patients' nutritional status and validated on Indian cancer patients.
Physical activity assessment (Indian Migrant Study Physical Activity questionnaire (IMS-PAQ) | 6 months
  Indian Migrant Study Physical Activity questionnaire (IMS-PAQ) was used to assess patients' physical activity throughout the day. We assessed physical activity at three time points during the study: baseline, at 3 months of intervention and at 6 months end of intervention.
  IMS-PAQ is a validated questionnaire on both Indian rural and urban population.
Quality of life (QoL) assessment (EORTC-QLQ- C30 questionnaire) | 6 months
  EORTC-QLQ- C30 questionnaire was used to analyse patients' QoL at baseline, mid- intervention and at the end of intervention period.
Haemoglobin (Haemoglobin levels) | 6 months
  Haemoglobin levels were monitored at baseline, at three months and at the end of intervention (6 months).
Serum albumin (Serum albumin levels) | 6 months
  Serum albumin levels were monitored at baseline, at three months and at the end of intervention (6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Ihab Tewfik, PhD, Principal Investigator — University of Westminster
Locations (2):
- All India Institute of Medical Sciences, New Delhi, India
- University of Westminster, London, United Kingdom

REFERENCES:
- [Derived] Kapoor N, Naufahu J, Tewfik S, Bhatnagar S, Garg R, Tewfik I. A Prospective Randomized Controlled Trial to Study the Impact of a Nutrition-Sensitive Intervention on Adult Women With Cancer Cachexia Undergoing Palliative Care in India. Integr Cancer Ther. 2017 Mar;16(1):74-84. doi: 10.1177/1534735416651968. Epub 2016 Jun 1. PMID 27252077